CLINICAL TRIAL: NCT02861209
Title: CONTACT: A Prospective Interventional Multicentre Before-after Study for the Implementation of a Care Pathway to Increase Self-management of Patients With Cancer Who Are Treated With Oral Anticancer Medications
Brief Title: Collaborative Network to Take Responsibility for Oral Anticancer Therapy
Acronym: CONTACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Lise-Marie Kinnaer, PharmD, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LMK15022016
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; ALL; Lung Cancer; Melanoma; Colorectal Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Melanoma; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-care pathway (No Intervention): This arm comprises patients before the implementation of the care pathway. Patients starting with an oral anticancer therapy participate in the current care process. Outcomes are assessed at start of treatment, after 1 and after 3 months.
  The decision to start with an oral anticancer therapy depends solely on the treating physician.
- Care Pathway (Experimental): This arm comprises patients after the implementation of the care pathway. Patients starting with an oral anticancer therapy in this arm, receive care as is described by the novel designed care pathway. Outcomes are again assessed at start of treatment, after 1 and after 3 months.
  The decision to start with an oral anticancer therapy depends solely on the treating physician.
  Interventions: Other: Implementation of a care pathway

INTERVENTIONS:
Other: Implementation of a care pathway — The care pathway will consist of procedures of care in the hospital (e.g. consultations with doctors, contact moments with nurses, ...) that describe the initiation of an oral anticancer therapy and the further follow up. The care pathway should describe how care can efficiently be organised.
  Arms: Care Pathway

SUMMARY:
This study aims to develop, implement and evaluate a care pathway for patients with cancer who are treated with oral anticancer drugs (OACD).

The care pathway will be developed in six hospitals in Flanders, and will be adapted to the local setting and situation.

The investigators hypothesize that the implementation of a care pathway will increase the quality of the drug therapy, the communication between health care professionals (HCPs) and patients, and will lead to an improved level of self-management and adherence. Moreover, the invesitgators hypothesize that the care pathway will facilitate the communication between HCPs in the hospital setting and in ambulatory care, and will improve counseling skills, self-efficacy and self-confidence of HCPs.

At the end of the study, a roadmap for the nation-wide implementation of a similar care pathway will be constructed based on the experiences of the participating hospitals. This roadmap will certainly include an e-learning platform for healthcare professionals.

DETAILED DESCRIPTION:
For each hospital, an individual care pathway will be developed following the 7-phase model by Vanhaecht et al., 2011. This methodology aims to offer a systematic approach in 7 phases for the support of an interdisciplinary team in the development of new care pathways or in the improvement of existing ones.

The before-part of the study includes phases 1 to 4 that aim to map current practice in detail and to translate these findings into the development of a care pathway. Current practice will be investigated using mixed methods comprising:

* surveys evaluating care on the level of the hospital
* semi-structured interviews with healthcare professionals (HCP) and patients
* outcome assessments in patients included in the study (self-management, adherence, satisfaction with care, satisfaction with information, quality of life) using validated questionnaires at the start of the therapy, after 1 month and after three months
* outcome assessments in healthcare professionals at baseline (self-efficacy and perceptions on self-management) using validated questionnaires
* training and feedback sessions on counseling for HCPs

Based upon these findings, a care pathway in each hospital will be developed by a local project team of different stakeholders from different disciplines.

The after-part of the study includes phase 5-7 in which the care pathway is implemented, evaluated and continuously followed up.

Implementation and evaluation take place at the same time. The evaluation includes:

* outcome assessments in patients (newly recruited) at the start of the therapy, after 1 month and after three months
* outcome assessments in HCPs (follow up)
* evaluation of counseling skills
* focus group discussions and interviews with HCPs to evaluate the development and implementation of the care pathway.

At the end of the study a comparison of outcomes before and after the implementation will be made to study the impact of the care pathway on the before mentioned aspects (see "Brief Summary").

ELIGIBILITY:
Inclusion Criteria:

* a hematological cancer of solid tumor
* starting an oral anticancer drug for the first time
* able to understand and speak Dutch

Exclusion Criteria:

* patients following an adjuvant oral anticancer therapy (e.g. tamoxifen)
* patients following a therapy with a study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Change in self-management skills | at the start of the therapy, after one and three months
  There is no gold standard to define self-management. A definition from Barlow et al., 2002 (2) defines self-management as follows: the ability of an individual to manage the symptoms, treatment, physical and psychosocial consequences and life style changes due to his/her condition. Adequate self-management refers to the ability to monitor one's condition and to effect cognitive, behavioural and emotional responses necessary to maintain a satisfactory quality of life.
  The studied self-management skills in this project comprise "social integration and support", "health service navigation", "constructive attitudes and approaches", "skill and technique acquisition" and "emotional distress".

SECONDARY OUTCOMES:
Change in medication Adherence | after one and three months of therapy
Change in patient satisfaction with treatment using the Cancer Therapy Satisfaction Questionnaire (CTSQ) | after one and three months
Change in patient satisfaction with care using Out-patsat 35 | at the start of the therapy, after one and three months
  The outpatsat is a questionnaire for ambulatory cancer patients in which they are asked to rate in different subscales their perceptions on care delivered by doctors, nurses and rate te overall organisation (accessibility of the hospital, ease of reaching the hospital by telephone, ...) during their stay at day hospital of consultations
Health Related Quality of Life | at the start of the therapy, after one and three months
Change in Distress using the Distress Barometer | at the start of the therapy, after one and three months
Efficacy of treatment Using ECOG performance scale and RECIST criteria | at the start of the therapy, after one and three months
Toxicity of treatment | at the start of the therapy, after one and three months
  Summarizing adverse drug events
Cost of care | at the start of the therapy, after one and three months
  Prospective report on health care expenditures (use of healthcare and other services, use of medicines, …)

OTHER OUTCOMES:
Change in Self-efficacy in HCPs using the Self-efficacy and Performance in Self-management Instrument (SEPSS) | at baseline (before the implementation of the care pathway) and after 24 months (during implementation)
  SEPSS investigates the ability of a HCP to evaluate their own performance in daily practice and caregiving.
Change in perceptions on self-management in HCPs using the Clinician Support for Patient activation measure | at baseline (before the implementation of the care pathway) and after 24 months (during implementation)

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - AZ Turnhout, Turnhout, Antwerpen
  - Maria Middelares Gent, Ghent, Oost-Vlaanderen
  - Imelda Bonheiden, Bonheiden, Vlaams-Brabant
  - AZ Groeninge Kortrijk, Kortrijk, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinnaer LM, Decoene E, Van Hecke A, Foulon V. Collaborative network to take responsibility for oral anticancer therapy (CONTACT): Study-protocol investigating the impact of a care pathway. J Adv Nurs. 2019 Dec;75(12):3726-3739. doi: 10.1111/jan.14157. Epub 2019 Aug 27. PMID 31310353